CLINICAL TRIAL: NCT04478565
Title: Development of Alternatives for the Estimation of the Resting Metabolic Rate From Anthropometric Variables in Paralympic Athletes
Brief Title: Development of Alternatives for the Estimation of the Resting Metabolic Rate From Anthropometry in Paralympic Athletes
Acronym: RMRPA
Status: Completed | Type: Observational
Sponsor: Iberoamerican Institute of Sports Science and Human Movement (Other)
Responsible Party: Principal Investigator, Cesar Octavio Ramos Garcia, PhD, Head of Research and Development, Iberoamerican Institute of Sports Science and Human Movement
Other Study IDs: IICDEM-ID-001-2020
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Resting Metabolic Rate; Disability Physical; Athletic Injuries
Keywords: Anthropometry; Indirect Calorimetry; Bioenergetics; Metabolic rate; Paralympic Athletes
MeSH Terms: conditions — Athletic Injuries | interventions — Calorimetry, Indirect; Anthropometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Indirect Calorimetry — RMR was calculated by breath oxygen consumption (O2 in mL·min-1), minute by minute, using a portable device (Breezing®, Arizona, USA), and the Weir equation (1949), while participants remained in a sitting position for ≈15 to 20 minutes.
  The anthropometric measurements were performed by certified level 3 anthropometrists following the guidelines of the International Society for the Advancement of Kinanthropometry, ISAK
  Other Names: Anthropometry

SUMMARY:
To our knowledge no study has evaluated neither feasible methods for the assessment of anthropometric profile nor indirect methods to estimate energy expenditure (EE) for adapted athletes. The primary aim is to develop and validate new RMR prediction models, for the estimation of the resting metabolic rate from anthropometric variables in young Mexican Paralympic athletes; our second objective is to evaluate the agreement between RMR and the prediction models of Cunningham, Harris-Benedict, Henry, Valencia, Chun, Nightingale & Gorgey, FAO/WHO, Mifflin, Müller, Owen, and our own models. A comparative cross-sectional quantitative study was designed. Participants report to the testing laboratory only once for data collection. The Strengthening the Reporting of Observational Studies in Epidemiology criteria guidelines for cross-sectional research (STROBE) is followed in the design/reporting of this study.

ELIGIBILITY:
Inclusion Criteria:

i) swimmers who report to the assessment area with a fasting period of 6 to 8 hours, and at least 12 hours after their last exercise routine; ii) swimmers who have not consumed alcohol or any stimulant for the last 48 hours (e.g., coffee, tea, chocolate, carbonated drinks, energy drinks, supplements); iii) swimmers who has contested at least in one of the last two swimming competitions, including World Championships and Paralympic Games

Exclusion Criteria:

i) fail to complete the indirect calorimetry test after two attempts; ii) attend to the evaluation area without the appropriate clothing or without following the instructions for fasting, exercise, and feeding prior to the evaluations; iii) swimmers who at the time of the evaluations did not give written consent (parental consent in case of under 18 years old) for procedures or data release for research purposes.

Ages: 10 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Mexican Paralympic swimmers from the national and the state adapted swimming team.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Indirect Calorimetry | One day
  The RMR was measured by IC using a portable device (Breezing®, Arizona, USA), which was calibrated before each test and has been described as a valid and reliable system (Xiaojun et al. 2015). RMR was calculated by breath oxygen consumption (O2 in mL·min-1), minute by minute, using the Weir equation (1949), while participants remained in a sitting position for ≈15 to 20 minutes.
Anthropometry | One day
  The anthropometric measurements were performed by certified level 3 anthropometrists following the guidelines of the International Society for the Advancement of Kinanthropometry, ISAK (Stewart et al, 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Alacid Cárceles, PhD, Principal Investigator — Universidad de Almeria; Luis A Quiroga Morales, PhD, Principal Investigator — Iberoamerican Institute of Sports Science and Human Movement; Diego A Bonilla Ocampo, PhD, Principal Investigator — DBSS International; Adrian J Martínez Rubio, MSc, Principal Investigator — Iberoamerican Institute of Sports Science and Human Movement
Locations (1):
- Iberoamerican Institute of Sports Science and Human Movement, Zapopan, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chun SM, Kim HR, Shin HI. Estimating the Basal metabolic rate from fat free mass in individuals with motor complete spinal cord injury. Spinal Cord. 2017 Sep;55(9):844-847. doi: 10.1038/sc.2017.53. Epub 2017 May 23. PMID 28534498
- [Result] Cunningham JJ. A reanalysis of the factors influencing basal metabolic rate in normal adults. Am J Clin Nutr. 1980 Nov;33(11):2372-4. doi: 10.1093/ajcn/33.11.2372. PMID 7435418
- [Result] Harris JA, Benedict FG. A Biometric Study of Human Basal Metabolism. Proc Natl Acad Sci U S A. 1918 Dec;4(12):370-3. doi: 10.1073/pnas.4.12.370. No abstract available. PMID 16576330
- [Result] Henry CJ. Basal metabolic rate studies in humans: measurement and development of new equations. Public Health Nutr. 2005 Oct;8(7A):1133-52. doi: 10.1079/phn2005801. PMID 16277825
- [Result] Mifflin MD, St Jeor ST, Hill LA, Scott BJ, Daugherty SA, Koh YO. A new predictive equation for resting energy expenditure in healthy individuals. Am J Clin Nutr. 1990 Feb;51(2):241-7. doi: 10.1093/ajcn/51.2.241. PMID 2305711
- [Result] Muller MJ, Bosy-Westphal A, Klaus S, Kreymann G, Luhrmann PM, Neuhauser-Berthold M, Noack R, Pirke KM, Platte P, Selberg O, Steiniger J. World Health Organization equations have shortcomings for predicting resting energy expenditure in persons from a modern, affluent population: generation of a new reference standard from a retrospective analysis of a German database of resting energy expenditure. Am J Clin Nutr. 2004 Nov;80(5):1379-90. doi: 10.1093/ajcn/80.5.1379. PMID 15531690
- [Result] Nightingale TE, Gorgey AS. Predicting Basal Metabolic Rate in Men with Motor Complete Spinal Cord Injury. Med Sci Sports Exerc. 2018 Jun;50(6):1305-1312. doi: 10.1249/MSS.0000000000001548. PMID 29315167
- [Result] Owen OE, Holup JL, D'Alessio DA, Craig ES, Polansky M, Smalley KJ, Kavle EC, Bushman MC, Owen LR, Mozzoli MA, et al. A reappraisal of the caloric requirements of men. Am J Clin Nutr. 1987 Dec;46(6):875-85. doi: 10.1093/ajcn/46.6.875. PMID 3687821
- [Result] WEIR JB. New methods for calculating metabolic rate with special reference to protein metabolism. J Physiol. 1949 Aug;109(1-2):1-9. doi: 10.1113/jphysiol.1949.sp004363. No abstract available. PMID 15394301